CLINICAL TRIAL: NCT06103487
Title: A Long-term Follow-up Study to Evaluate the Safety of RGX-111
Brief Title: Long Term Follow-Up for RGX-111
Status: Enrolling by invitation | Type: Observational
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-111-5101
Record Dates: First submitted 2023-10-05; First posted 2023-10-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Mucopolysaccharidosis I
Keywords: MPS I; hurler syndrome; gene therapy
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RGX-111 Recipients: Subjects who have received RGX-111 in a separate parent study.
  Interventions: Genetic: No Intervention

INTERVENTIONS:
Genetic: No Intervention — Observational study

SUMMARY:
RGX-111-5101 is a long-term follow up study that evaluates the long term safety of RGX-111 in participants who have received RGX-111 (a gene therapy intended to deliver a functional copy of the alpha-L-iduronidase gene (IDUA) to the central nervous system) in a separate parent study.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational, follow-up study to evaluate the long-term safety of RGX-111 after a single administration. Eligible participants are those who previously participated in a clinical study where they received a single IC or ICV administration of RGX-111. Enrollment of each participant in this study should occur on the same day or after the participant has completed the end of study (EOS) visit or early discontinuation visit (EDV) from a previous (parent) clinical study. Participants will be followed for up to five years after RGX-111 administration (inclusive of the parent study) or until RGX-111 is commercially available in the participant's country, whichever occurs first. No treatment will be directed under this observational protocol. The total study duration for each participant may vary depending on when s/he enrolls in the current study following RGX-111 administration in the parent study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, a participant must have previously received RGX-111 in a separate parent trial.
* Participant or participant's legal guardian(s) is/(are) willing and able to provide written, signed informed consent.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Received RGX-111 in a separate parent trial.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the long-term safety of RGX-111 | 5 years inclusive of parent study
  Incidences of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) over time

SECONDARY OUTCOMES:
Safety and Efficacy: Change from baseline in neurodevelopmental parameters | 5 years inclusive of parent study
  Change in baseline adaptive behavior as measured by Vineland Adaptive Behavior Scales Third Edition (VABS-III). The VABS-III assesses adaptive behavior in individuals from infancy to age 90 years. In this study, 4 domains of Communication, Daily Living Skills, Socialization, and Motor Skills will be assessed. The domains have different scoring ranges, with higher subdomain raw scores indicating greater function, but can be normalized for cross-domain comparison.

CONTACTS AND LOCATIONS:
Locations (2):
- Children's Hospital of Orange County, Orange, California, United States
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No